CLINICAL TRIAL: NCT01379053
Title: Detection of Methicillin Resistant Staphylococcus Aureus Colonization Using the zNose®, an Ultra-fast Gas Chromatograph
Brief Title: Volatile Organic Compounds in Staphylococcus Aureus Patients
Acronym: MRSAVOC
Status: Completed | Type: Observational
Sponsor: Landon Pediatric Foundation (Other)
Responsible Party: Principal Investigator, Chris Landon, Principal Investigator, Landon Pediatric Foundation
Other Study IDs: MRSA1
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Staphylococcus Aureus; Methicillin-resistant Staphylococcus Aureus; Nosocomial Disease
Keywords: Staphylococcus aureus; Methicillin-resistant staphylococcus aureus; Nosocomial disease; Electronic nose; Gas chromatography
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Staphylococcus Patients: Patients suspected of having Methicillin-resistant and/or methicillin-susceptible staphylococcus aureus.
- Control: Healthy volunteer

SUMMARY:
The zNose® MRSA test is a non-invasive breath test for markers of Staphylococcus aureus, which may predict the probability of bacterial organisms in the anterior nares, throat and respiratory tract, wounds, and anus and therefore be able to replace or supplement current active Methicillin Resistant Staphylococcus Aureus (MRSA) surveillance efforts. It consists of:

* A collection apparatus for collection of volatile compounds from suspected infection sites onto a sorbent trap or Tedlar bag, as well as for the collection of a separate sample of room air.
* Analysis of the volatile organic compounds from suspected infection sites and room air by short acoustic wave gas chromatography.
* Interpretation of the volatile organic compounds with a proprietary algorithm in order to predict the probability of Staphylococcus aureus infection and colonization.

This study will test the hypothesis that we can identify the presence of MRSA by sampling the "head space" above culture media of anterior nare samples provided by patients with MRSA. Additionally, this study will test the hypothesis that we can identify the presence of MRSA by sampling air exhaled through the nostrils (nasal exhalant).

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of staphylococcus aureus infection or colonization
* Able to give samples for zNose® analysis

Exclusion Criteria:

* Inability to provide sample for zNose® analysis

Ages: 1 Year to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be selected upon suspicion of MRSA or MSSA infection or colonization. Increased concentration will be give to selection of persons from the following high risk groups:
  * It has been documented that the patient has been previously discharged from a general acute care hospital within 30 days prior to the current hospital admission.
  * The patient will be admitted to an intensive care unit or burn unit of the hospital.
  * The patient receives inpatient dialysis treatment.
  * The patient is being transferred from a skilled nursing facility
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Identification of Methicillin Resistant Staphyloccus aureus | one week
  Identification during clinic visit of MRSA

CONTACTS AND LOCATIONS:
Locations (1):
- Ventura County Medical Center Hospital, Ventura, California, United States